CLINICAL TRIAL: NCT05546216
Title: Determination of the Effect of Raised Supine Position and Back Support on Back Pain, Anxiety and Comfort Level in Coronary Angiography Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, AYSE SOYLU, Lecturer, Doctor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: İnönü
Record Dates: First submitted 2022-09-16; First posted 2022-09-19 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Coronary Angiography Patient; Anxiety; Back Pain; Comfort
Keywords: Patient Position; Pillow
MeSH Terms: conditions — Anxiety Disorders; Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patients in the intervention group CAG exit Written informed consent was obtained from the patients for the study. Pretest data of the patients were collected at 0 hour using the "Patient Information Form", "Visual Analog Scale", "State Anxiety Scale" and "Immobility Comfort Scale". After informing the patient with hemodynamics, at the 0th hour, a 36x33x10 cm gel-containing silicone pad was placed in the lumbar cavity of the patient to fill the patient's anatomical lumbar cavity, and CAG output was supported. The patient was in the supine position 30 degrees elevated when measured with the visual aid. Patients lie in the same position for 4 hours. Back pain of the patients was evaluated again with the "Visual Analog Scale" at the 2nd hour. At the 4th hour, the posttest data of the patients were collected with the "Visual Analogue Scale", the "State Anxiety Scale" and the "Immobility Comfort Scale".
  Interventions: Other: Determination of the Effect of Raised Supine Position and Back Support on Back Pain, Anxiety and Comfort Level in Coronary Angiography Patients
- control group (No Intervention): After the patients in the control group were placed in the supine position on the CAG exit, they were monitored, their vital signs were evaluated, and the necessary information of the patient was collected with the "Patient Information Form", "Visual Analog Scale", "State Anxiety Scale" and "Immobilization comfort scale" at the 0th hour of CAG exit. The patient was in a routine supine position without back support for 4 hours and received standard nursing care. After the . position was given, back pain was evaluated again at the 2nd hour and 4th hour using the "Visual Analogue Scale". Anxiety and comfort levels were evaluated with the "State Anxiety Scale" and "Immobilization Comfort Scale" at the 0th minute before the position and at the 4th hour after the position .

INTERVENTIONS:
Other: Determination of the Effect of Raised Supine Position and Back Support on Back Pain, Anxiety and Comfort Level in Coronary Angiography Patients — The study was conducted between 01 September 2021 and 30 January 2022 as a randomized single-blind interventional study with a pre-test post-test control group. The sample of the study consisted of patients who underwent coronary angiography. Data; The patient information form was collected with the visual analog scale, state anxiety and immobilization comfort scale. Back support was provided to the intervention group with a pillow at the exit of the angiography and the head of the bed was raised 30 degrees. Back pain intensity at 0, 2 and 4 hours, anxiety and comfort level at 0 and 4 hours were measured. The control group was given routine nursing care.
  Arms: Experimental group

SUMMARY:
In addition to pharmacological methods, non-pharmacological methods are also used to control back pain and anxiety. The aim of the study is to determine the effect of 30 degrees raised supine position and back support applied to patients undergoing coronary angiography from the femoral artery on back pain, anxiety and patient comfort. This research was planned as a pretest-posttest randomized, controlled, experimental study in order to determine the effect of the elevated supine position and back support application applied to patients undergoing coronary angiography with femoral artery access on back pain, anxiety and comfort levels of patients.

Research Kahramanmaraş Sütçü İmam University SUAH Hospital Cardiology intensive care unit September 2021 - September The sample of the research was determined by power analysis. According to the calculation made, the sample; With an effect size of 0.90, a margin of error of 0.05, a confidence interval of 0.95, and a power of 0.95, it was calculated that there should be 35 people in each group to represent the universe. "Patient Information Form", "Numeric Pain Intensity Scale VAS", "State- The necessary information of the patient will be collected with the "Trait Anxiety Scale" and the "Immobilization comfort scale". After the information of the patient whose hemodynamics is provided, the experimental group will be given a 30 degrees Elevated Supine Position and the back area will be supported with a 36x33x10 sized silicone gel pad that prevents sweating, and the measurements will be repeated at the 2nd and 4th hours after the CAG procedure.

The patients in the control group will have the same measurements at the 0th hour, 2nd hour and 4th hour after the femoral angiography procedure. During this period, the patients will remain in the straight supine position without back support, which is routinely applied in the clinic.

DETAILED DESCRIPTION:
Coronary Artery Disease (CAD) is the most common system disease among cardiovascular system diseases (CVS). CVS diseases are in the first place among the top 10 causes of death stated by the World Health Organization (WHO). Every year, 17.9 million people in the world die due to CVS diseases. A similar picture is seen in our country with the world average, and according to the 2013 data of the Turkish statistical institution, 37.9% of all deaths are due to CAD. In the heart disease risk factor study of Turkish adults in 2017, the death rate of CAD in European countries between the ages of 45-74 is between 2 and 8 per thousand in men and between 0.6 and 3 per thousand in women. This rate has been reported as 7.6 in men and 3.8 in women between the ages of 45-74 in our country. Coronary angiography (CAG) procedure is currently the gold standard in the diagnosis and treatment of CAD. Complications such as bleeding, hematoma and arterial embolism may develop after CAG. Complete bed rest is recommended for approximately 6 hours after CAG to minimize these risks. During bed rest, the patient lies motionless in the supine position. Studies in the literature have also reported that lying still after CAG causes back pain. Back pain after CAG may increase sympathetic stimulation. Therefore, heart rate, blood pressure, myocardial oxygen consumption and cardiac workload increase. This may exacerbate myocardial ischemia. It is also reported in the literature that CAG is a cause of anxiety for patients. In patients hospitalized in the coronary intensive care unit after the procedure, the presence of anxiety reduces the quality of life and increases the frequency of acute coronary events, and may lead to increased mortality. In addition to pharmacological methods, non-pharmacological methods are also used to control back pain and anxiety. The aim of the study is to determine the effect of 15 degrees raised supine position and back support applied to patients undergoing coronary angiography from the femoral artery on back pain, anxiety and patient comfort. This research was planned as a pretest-posttest randomized, controlled, experimental study in order to determine the effect of the elevated supine position and back support application applied to patients undergoing coronary angiography with femoral artery access on back pain, anxiety and comfort levels of patients.

The research will be carried out in Kahramanmaraş Sütçü İmam University SUAH Hospital Cardiology intensive care unit between September 2021 and September 2022.

There is an annual average of 436 patients hospitalized for CAG in the Coronary intensive care unit in the relevant hospital. The sample of the study was determined by power analysis. According to the calculation made, the sample; With an effect size of 0.90, a margin of error of 0.05, a confidence interval of 0.95, and a power of 0.95, it was calculated that there should be 35 people in each group to represent the universe. However, considering the losses that may be experienced during the study, it was decided that it would be appropriate to take 10 extra people and each group was planned as 45 people (45+45 Experimental-Control Group). It was aimed to reach 90 patients in total. Volunteers aged 18 and over, who do not have communication barriers that may affect cognitive functions, and patients who underwent femoral angiography will be randomly assigned to the study. Data will be collected using face-to-face interview method.

The data of the study were collected from the "Patient Information Form", "Numeric Pain Intensity Scale", "State Anxiety Scale", "Immobilization comfort scale", "Back support and 15 degrees Elevated Supine Position practice plan.

The patients in the experimental group will be monitored after they are put to bed after the angiography procedure, their vital signs will be evaluated at the 0th hour, "Patient Information Form", "Numeric Pain Intensity Scale VAS (Numeric Pain Intensity Scale)", "State-Trait Anxiety Scale" and "Immobilization Comfort Scale". The necessary information of the patient will be collected with the "scale". After the information of the patient whose hemodynamics is provided, the experimental group will be given a 15 degree Elevated Supine Position and the back area will be supported with a 36x33x10 sized silicone gel pad that prevents sweating, and the measurements will be repeated at the 2nd and 4th hours after the CAG procedure.

The patients in the control group will have the same measurements at the 0th hour, 2nd hour and 4th hour after the femoral angiography procedure. During this period, the patients will remain in the straight supine position without back support, which is routinely applied in the clinic.

ELIGIBILITY:
Inclusion Criteria:

* No communication barrier that will affect cognitive functions, 18 years old and over, Femoral angiography procedure performed.

Exclusion Criteria:

* Bilinci kapalı olan, Psikiyatrik bir hastalığı olan, Sırt ameliyatı geçiren/bel fıtığı olan, Kronik bel veya sırt ağrısı olan, Radiyal anjiyografi işlemi yapılan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Back pain | 4 hour
  The patient will also have less back pain.
Anxiety | 4 hour
  Patient anxiety will decrease
Comfort | 4 hour
  Patient comfort will increase

CONTACTS AND LOCATIONS:
Locations (1):
- KahramanmarasSIU, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual data will be kept confidential

REFERENCES:
- [Derived] Soylu A, Korkmaz M. The effect on back pain, anxiety, and comfort levels of an elevated supine position and back support applied to patients undergoing coronary angiography: A randomized controlled experimental study. Saudi Med J. 2024 Jul;45(7):700-709. doi: 10.15537/smj.2024.45.7.20240201. PMID 38955437
- Available data/document: REFERENCE — https://doi.org/10.1016/j.ctcp.2019.101068
- Available data/document: REFERENCE — http://dx.doi.org/10.1016/j.ijcard.2016.11.043
- Available data/document: REFERENCE — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4540812/
- Available data/document: REFERENCE — https://pubmed.ncbi.nlm.nih.gov/30367542/
- Available data/document: REFERENCE — https://pubmed.ncbi.nlm.nih.gov/18065335/
- Available data/document: REFERENCE — https://pubmed.ncbi.nlm.nih.gov/35307131/
- Available data/document: REFERENCE — https://pubmed.ncbi.nlm.nih.gov/17056770/
- Available data/document: REFERENCE — https://pubmed.ncbi.nlm.nih.gov/27252099/
- Available data/document: REFERENCE — https://pubmed.ncbi.nlm.nih.gov/33632127/
- Available data/document: REFERENCE — https://pubmed.ncbi.nlm.nih.gov/26171374/
- Available data/document: REFERENCE — https://pubmed.ncbi.nlm.nih.gov/29476940/